CLINICAL TRIAL: NCT02398747
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AZD2014 Administered to Japanese Patients With Advanced Solid Malignancies
Brief Title: Japanese Phase I Study of AZD2014 in Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2270C00008
Record Dates: First submitted 2015-03-10; First posted 2015-03-25 (Estimated); Last update posted 2024-12-17 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Malignancies
MeSH Terms: interventions — vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD2014 50mg, 125mg, 25mg and 50mg intermittent BD (Experimental): 50mg BD continuous dosing, 125mg BD intermittent dosing, 25 mg and 50mg intermittent dosing with weekly Paclitaxel
  Interventions: Drug: AZD2014

INTERVENTIONS:
Drug: AZD2014 — 50mg continuous dosing, 125mg intermittent dosing, 25 mg and 50mg intermittent dosing with weekly Paclitaxel

SUMMARY:
The primary objective of this study is to investigate the safety and tolerability of continuous and/or intermittent dosing of AZD2014 when given orally to patients with advanced solid malignancies.

DETAILED DESCRIPTION:
This is an open-label, multi-centre study of AZD2014 administered orally in Japanese patients with advanced solid malignancies. The study design allows an evaluation of each cohort with intensive safety monitoring to ensure the safety of the patients. In this study, a minimum of 3 and a maximum of 6 evaluable patients will be enrolled in each cohort; approximately 24 evaluable patients in total. The total number of patients enrolled will depend upon the number of screen failures, number of cohorts and number of evaluable subjects.

Safety, preliminary efficacy and PK (single and multiple dose) are evaluated in this study.

Patients will receive a single dose of AZD2014 on Day 1 (to allow assessment of single dose PK), then after a minimum of 48 hours washout period continuous or intermittent twice daily dosing of AZD2014 will be initiated. The washout period of 48 hours may be extended depending on emerging data from previous cohorts.Doses and schedules to be evaluated will be agreed by AstraZeneca and the Safety Review Committee (SRC).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of a solid, malignant tumour that is refractory to standard therapies or for which no standard therapies exist
* For Cohort 3-1 and 3-2, followed as, Histological or cytological confirmation of a solid, malignant tumour that is refractory to standard therapies or for which no standard therapies exist or where treatment with paclitaxel is an appropriate treatment option. SqNSCLC patients are excluded from the Cohort 3-2.
* World Health Organisation (WHO) performance status (PS) 0-1 with no deterioration over the previous 2 weeks prior to informed consent and minimum life expectancy of 12 weeks
* At least one lesion that can be accurately assessed at baseline by computed tomography (CT) magnetic resonance imaging (MRI) or plain X-ray and is suitable for repeated assessment

Exclusion Criteria

* Prior chemotherapy, biological therapy, radiation therapy, antiandrogens, other anticancer therapies including immunotherapy and any investigational agents within 21 days of starting study treatment (not including palliative radiotherapy at focal sites), or corticosteroids within 14 days of starting study treatment.
* Major surgery within 4 weeks prior to the study treatment (excluding placement of vascular access), or minor surgery within 2 weeks prior to the study treatment
* Potent or moderate inhibitors or inducers of cytochrome (CYP) 3A4/5 if taken within the stated washout periods:
* Potent or moderate inhibitors or inducers of CYP2C8 if taken within the stated washout periods:
* Exposure to sensitive or narrow therapeutic range substrates of the drug metabolising enzymes CYP2C8, CYP2C9, CYP2C19, CYP2D6 or the drug transporters P-gp (MDR1), Breast cancer resistance protein (BCRP), Organic anion transporting polypeptide (OATP)1B1, OATP1B3, Organic cation transporter (OCT)1 and OCT2 within the appropriate wash-out period (at least 5 x reported terminal elimination half-life (t1/2) of each drug) before the study treatment.
* Any haemopoietic growth factors (eg, granulocyte-colony stimulating factor [G-CSF]) within 2 weeks prior to receiving study drug
* Previous initiation of treatment with AZD2014 in the present study or prior treatment with AZD8055
* With the exception of alopecia, any unresolved toxicities from prior chemotherapy greater than Common toxicity criteria for adverse events (CTCAE) grade 1 at the time of starting study treatment
* Spinal cord or brain metastases unless asymptomatic and stable off steroids for at least 4 weeks prior to start of study treatment
* Subjects with interstitial lung disease as a complication or a history

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured by adverse events | 6 months in average
  This will be assessed in terms of Adverse Events (AEs), laboratory data, vital signs, ECG and physical exams

SECONDARY OUTCOMES:
Cmax of AZd2014 | 21 days
  Characterising the pharmacokinetics (PK) of AZD2014
AUC(Area under the plasma concentration-time curve) of AZD2014 | 21 days
  Characterising the pharmacokinetics (PK) of AZD2014
Tmax of AZD2014 | 21 days
  Characterising the pharmacokinetics (PK) of AZD2014
To obtain a preliminary assessment of the anti-tumour activity of AZD2014 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. | 6 months in average
  Best overall response
To obtain a preliminary assessment of the anti-tumour activity of AZD2014 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. | 6 months in average
  Objective response rate
To obtain a preliminary assessment of the anti-tumour activity of AZD2014 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. | 6 months in average
  Percentage change in tumour size

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: AstraZenecaClinicaltrials.com — https://www.astrazenecaclinicaltrials.com/study/D2270C00008/